CLINICAL TRIAL: NCT05952505
Title: Immunogenicity and Safety of an Inactivated SARS-CoV-2 Vaccine Coadministered With Varicella Vaccine and Measles, Mumps and Rubella Combined Vaccine in Shanghai, China: A Non-inferiority, Open-label, Randomised, Controlled, Phase 4 Trial
Brief Title: Immunogenicity and Safety of an Inactivated SARS-CoV-2 Vaccine Coadministered With Two Attenuated Vaccines
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Municipal Center for Disease Control and Prevention (Other)
Collaborators: China National Biotec Group Company Limited (Industry)
Responsible Party: Principal Investigator, HUANG Zhuoying, Doctor, Shanghai Municipal Center for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SH2023-9
Record Dates: First submitted 2023-07-17; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV-2 Infection; Varicella; Measles; Mumps; Rubella
Keywords: Inactivated SARS-CoV-2 vaccine; coadministeration; varicella vaccine; measles, mumps and rubella combined vaccine
MeSH Terms: conditions — COVID-19; Chickenpox; Measles; Mumps; Rubella

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): immunized inactivated SARS-CoV-2 vaccine and varicella vaccine in day 0 followed by measles-mumps-rubella vaccine(MMR) in day 28.
  Interventions: Biological: Inactivated SARS-CoV-2 vaccine coadministered with vricella vaccine
- Group 2 (Experimental): immunized varicella vaccine in day 0 followed by SARS-CoV-2 vaccine and MMR in day 28.
  Interventions: Biological: Inactivated SARS-CoV-2 vaccine coadministered with MMR
- Group 3 (Active Comparator): immunized inactivated SARS-CoV-2 vaccine in day 0 followed by MMR and varicella vaccine in day 28.
  Interventions: Biological: Inactivated SARS-CoV-2 vaccine administered alone

INTERVENTIONS:
Biological: Inactivated SARS-CoV-2 vaccine coadministered with vricella vaccine — Subjects will be coadministered with inactivated SARS-CoV-2 vaccine and varicella vaccine.
  Arms: Group 1
Biological: Inactivated SARS-CoV-2 vaccine coadministered with MMR — Subjects will be coadministered with SARS-CoV-2 vaccine and MMR.
  Arms: Group 2
Biological: Inactivated SARS-CoV-2 vaccine administered alone — Subjects will be immunized with inactivated SARS-CoV-2 vaccine alone
  Arms: Group 3

SUMMARY:
Eligible participants were randomly assigned (1:1:1), using block randomization stratified, to either 3 groups. Group 1 will be immunized inactivated SARS-CoV-2 vaccine and varicella vaccine in day 0 followed by measles-mumps-rubella vaccine(MMR) in day 28.

Group 2 will be immunized varicella vaccine in day 0 followed by SARS-CoV-2 vaccine and MMR in day 28.

Group 3 will be immunized inactivated SARS-CoV-2 vaccine in day 0 followed by MMR and varicella vaccine in day 28.

Vaccines were administered 28 days apart, with blood samples taken on day 0 and day 28 before vaccination, and on day 56. Local and systemic symptoms and serious adverse events following immunzation were collected.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 years old
* With legal guardian signing the informed consent
* Able to participate in all planned visits and comply with all research procedures (such as completing diary cards of adverse events and participating visits)
* With clear vaccination records including no SARS-CoV-2 vaccine history, with 1 varicella vaccine and 2 measles-containing vaccines history
* the last attenuated vaccine was administered ≥28 days ago, and other vaccines administered ≥14 days ago
* With an axillary temperature ≤37.5℃ at the time of vaccination

Exclusion Criteria:

First dose exclusion criteria:

* With SARS-CoV-2 infection in the last 3 months (any of the following conditions shall be met: positive nucleic acid test; positive antigen test; suspected SARS-CoV-2 infection symptoms of subject or close contacts)
* allergic to any substance of the vaccine or with a severe allergic reactions history of vaccines (such as acute allergic reactions, angioneurotic edema, breathing difficulties, etc.)
* Suffering uncontrolled epilepsy or progressive nerve system diseases, or with a history of Gribali syndrome
* With acute illness, severe or acute attack of chronic illness or fever
* With immunodeficiency or weakened immune system or being treated with immunosuppressant drugs (oral steroids)
* Received non specific immunoglobulin within 3 months
* Any situation that researchers thought that might influence the consequence of the clinical trial Second dose exclusion criteria：
* Occurrence of any serious adverse event that may be related to the previous dose of study vaccine
* Occurrence of systemic adverse reactions or allergic reactions with a severity level ≥ 3 recognized by researchers after vaccination
* Any new situations that fit the first dose exclusion criteria
* Any situation that researchers thought that might influence the consequence of the clinical trial

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
non-inferiority of the seroconversion rate and neutralising antibody level against SARS-CoV-2 | on day 28 after vaccination
  Neutralizing antibody of SARS-CoV-2 is an index of immunogenicity
non-inferiority of the seroconversion rate and IgG antibody level against measles, rubella, and mumps | on day 28 after vaccination
  IgG antibodies of measles, rubella, and mumps is an index of immunogenicity
non-inferiority of the seroconversion rate and IgG antibody level against varicella | on day 28 after vaccination
  IgG antibodies of varicella is an index of immunogenicity

SECONDARY OUTCOMES:
incidence of reported vaccine-related adverse events within 28 days of each immunization. | from 0 to 28 days after vaccination
  adverse events including local and systemic symptoms followng immunization

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoying Huang, Study Director — Shanghai Municipal Center for Disease Control and Prevention
Locations (1):
- Shanghai Municipal Center for Disease Control and Prevention, Shanghai, Shanghai Municipality, China